CLINICAL TRIAL: NCT04214704
Title: Assessing the Benefits of a Painless Lancing Device Among Diabetes Subjects in Improving Self-monitoring Frequency and HbA1c
Brief Title: Assessing the Benefits of a Painless Lancing Device Among Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jothydev's Diabetes and Research Centre (Other)
Responsible Party: Principal Investigator, Dr. Jothydev Kesavadev, Chief Diabetologist and Chairman, Jothydev's Diabetes and Research Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JDC/GENTEEL/022/2019
Record Dates: First submitted 2019-12-27; First posted 2020-01-02 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: lancing device; HbA1c; painless lancing; SMBG adherence
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Genteel arm (Experimental): In the Genteel arm, the subjects exclusively use the Genteel device for the first 12 weeks, and then switch to the conventional method of SMBG for an additional 12 weeks. This arm will use Butterfly Touch Lancets (BTL) throughout the study.
  Interventions: Device: Genteel lancing device; Device: Conventional lancing device
- Conventional arm (Active Comparator): In the Conventional arm, the subjects use the conventional method of SMBG for the first 12 weeks and then switch to the Genteel device for an additional 12 weeks. This arm will use the lancet and lancing device which they were using prior to randomization to the study.
  Interventions: Device: Genteel lancing device; Device: Conventional lancing device

INTERVENTIONS:
Device: Genteel lancing device — Painless lancing device that helps to improve and assess self-monitoring frequency and HbA1c respectively
Device: Conventional lancing device — Conventional lancing device

SUMMARY:
The purpose of this study is to assess the benefits of a painless lancing device among diabetes subjects in improving self-monitoring frequency and HbA1c compared to the conventional lancing device.

DETAILED DESCRIPTION:
Self-monitoring of glucose forms the cornerstone of diabetes management. There are multiple limiting factors towards efficient self- monitoring of blood glucose, including cost barriers, inconvenience, investment of time, pain associated with pricking etc. Pain has perceived as a major impediment to the self-monitoring of blood glucose.

Genteel lancing device offers a painless pricking experience and hence helps to report blood sugar values at least 4 times a day. The perceived pain sensitivity of the study subjects would be assessed using the 4- point pain screening questionnaire during the course of the study.

The aim of this study is to gather information on the percentage reduction in HbA1c values in diabetes patients as compared to the baseline values after three months and six months respectively brought about by percentage SMBG adherence, defined as the percentage of total recorded SMBG values as compared to the ideal number of readings over the 24-week period. SMBG adherence = actual number of fingerpricks (6 times daily in type 1 subjects or twice weekly in type 2 subjects).

SMBG adherence can be provisionally attained by multiple pricking using painless Genteel lancing device compared to the conventional lancing device. Additionally, the subject is asked about the likelihood they would use the device if available for routine SMBG practice in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Less than or equal to 70 years of age. If minor (<18 years), accompanied by caretaker.
2. Diagnosed with either Type 1 or Type 2 diabetes including newly diagnosed. 50% of the study participants will be type 1 diabetes subjects and 50% will be type 2 diabetes subjects
3. Presenting with an uncontrolled glycemic status (HbA1c >8.0%).
4. Ready for Self-Monitoring of Blood Glucose (SMBG) practices.
5. Attending physician prescribed testing at least 2 times per day
6. Judged by the study trainer to be competent to correctly use Genteel AND demonstrated to the trainer that the subject can use the Genteel device properly.

Exclusion Criteria:

1. More than 70 years and less than 5 years
2. HbA1c < 8.0%
3. Unwilling for SMBG.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Percentage SMBG adherence | 24 weeks
  Percentage SMBG adherence, defined as the percentage of total recorded SMBG values as compared to the ideal number of readings over the 24-week period.SMBG adherence = actual number of fingerpricks/ ideal number of fingerpricks(6 times daily in type 1 subjects or twice weekly in type 2 subjects). Should be assessed both at baseline and end of 24 weeks.
Percentage reduction in HbA1c | 24 weeks
  2) Percentage reduction in the HbA1c values as compared to the baseline values at 12 weeks and 24 weeks.

SECONDARY OUTCOMES:
Subjective assessment of pain reduction after using Genteel | 24 weeks
  The subject's Subjective Assessment of pain after using the Genteel device in comparison to conventional SMBG devices would be recorded using a pain scale.
  The scale for pain sensation is as follows:
  1. Elimination
  2. Significant reduction
  3. Slight reduction
  4. No change
  5. Mild worsening of pain
  6. Significant worsening of pain
  The above values are computed relative to the worst pain the subject can think of at a score of 6.
Subjective assessment of probability of using Genteel for SMBG | 24 weeks
  The subject is asked about the likelihood they would use the device if available for routine SMBG practices in the future. Scale for predicting future (probability) use of device for SMBG is as follows:
  1. Definitely yes
  2. Probably yes
  3. Not sure
  4. Probably no
  5. Definitely no
  The above values are computed relative to the worst probability this device would not be used in future at a score of 5.

CONTACTS AND LOCATIONS:
Overall Officials: Jothydev Kesavadev, MD, Principal Investigator — Jothydev's Diabetes Research Center
Locations (1):
- Jothydev's Diabetes Research Center, Trivandrum, Kerala, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] R. Warrier, S. Badarudeen, A. Shankar, G. Krishnan, L. Ramachandran, K. Thampiraj, S. Jothydev, J. Kesavadev. Assessing the Benefits of a Painless Lancing Device in a Subset of Patients Fearful of Finger Pricking. Diabetes Technol Ther. 2019. 21. A60-A61.